CLINICAL TRIAL: NCT04940780
Title: Examining the Impact of an Integrative Oncology Program on Patient Symptoms and Quality of Life: a Prospective Pragmatic Registry Protocol Study
Brief Title: Integrative Oncology for Patient Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Noah Samuels, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTEGR.ONCOL.REGIST-2021
Record Dates: First submitted 2021-06-16; First posted 2021-06-28 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Oncologic Complications; Symptoms and Signs
Keywords: Integrative medicine; Integrative oncology; Acupuncture; Touch therapy; Wellbeing
MeSH Terms: conditions — Signs and Symptoms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Patient-preference, pragmatic methodology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Preference Arm (Active Comparator): patients who specify their preference for either acupuncture or touch therapy
  Interventions: Other: Acupuncture; Other: Touch Therapies
- Randomized Treatment Arm (Active Comparator): with no preference, to be randomly allocated to either the acupuncture or touch-therapy subgroup
  Interventions: Other: Acupuncture; Other: Touch Therapies

INTERVENTIONS:
Other: Acupuncture — Acupuncture points will be selected on an individualized and symptom-directed basis, with the incorporation of points shown in clinical research to be effective for specific symptoms
Other: Touch Therapies — Touch therapies are to include Reflexology, Shiatsu and Therapeutic Touch

SUMMARY:
The use of complementary and integrative medicine (CIM) among oncology patients is widespread, with a large body of research-based evidence supporting the ability of these therapies to alleviate symptoms related to cancer and its treatment. Organizations such as the American Society for Clinical Oncology and the European Society for Medical Oncology have included CIM modalities in their treatment guidelines, and many of today's leading cancer centers include CIM in their supportive care service. The proposed study will prospectively examine the impact of a CIM treatment program on the symptom burden, quality of life and function of patients undergoing active oncology treatment.

A total of 750 patients will undergo an integrative oncologist (IP) consultation followed by a series of 8 CIM treatments consisting of either acupuncture or touch-related therapies (reflexology, Shiatsu, Tuina, etc.) with the goal of relieving their symptoms. Patients will be allocated to one of the two study treatment arms: the "Patient-Preference Arm", for patients who specify their preference for either acupuncture or touch therapy; and the "Randomized Treatment Arm", for those with no preference, to be randomly allocated to either the acupuncture or touch-therapy subgroup. Patients will be asked to complete the following study questionnaires before and after the treatment regimen: the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30); the Edmonton Symptom Assessment System (ESAS); and the Measure Yourself Concerns and Wellbeing (MYCAW) tool. The primary study outcome will be the change in EORTC Global Health-Status / Quality of Life scores, from pre- to post-treatment. Secondary study outcomes will include EORTC QLQ-C30 functional and symptom scales, single items assessing additional symptoms commonly reported by cancer patients, and perceived financial impact of the disease; ESAS severity scores for 10 quality-of life related items; and MYCAW severity scores for the 2 most significant symptoms, as well as post-treatment narratives. Other secondary outcomes to be assessed include the safety of the study treatments (adverse effects); adherence to conventional treatment regimen; and narratives from the patient's informal caregiver (spouse, parent/child, sibling, friend, etc.).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* undergoing active oncology treatment
* fully understand the study plan
* agree to sign the study informed consent form.

Exclusion Criteria:

* not fulfilling all of the study criteria
* not interested in attending all 8 weekly CIM treatments sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 global health status / QoL scale | 8 weeks
  Change from baseline to the end of the 8-week integrative treatment program

SECONDARY OUTCOMES:
EORTC QLQ-C30 global health status / QoL scale | 16 weeks
  Change from baseline and 8-week assessment to 16 week follow-up
EORTC QLQ-C30 - additional outcomes | From baseline to 8- (end of treatment program) and 16-week (post-program) assessment
  Change in functional and symptom scores
ESAS symptom severity scores | From baseline to 8- (end of treatment program) and 16-week (post-program) assessment
  Change in severity scores for 10 quality-of life related items
MYCAW symptom severity scores | From baseline to 8- (end of treatment program) and 16-week (post-program) assessment
  Change in severity scores for the 2 most significant symptoms, as well as post-treatment narratives
Frequency of adverse effects | At the end of the series of 8 weekly CIM treatment sessions (≤ 2 weeks after the last treatment session); after 16 weeks from baseline.
  Any reported adverse events taking place during the study period which are considered to have possibly/probably resulted from the CIM intervention
Adherence to conventional oncology treatment regimen | At 16 weeks from baseline.
  Adherence to oncology treatment to be measured using the Relative Dose Intensity (RDI) calculation
Caregiver expectations | At baseline
  Narratives from the patient's informal caregiver (spouse, parent/child, sibling, friend, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology, Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samuels N, Oberbaum M, Ben-Arye E. Expectations of Patients and Their Informal Caregivers from an Integrative Oncology Consultation. Integr Cancer Ther. 2021 Jan-Dec;20:1534735421990080. doi: 10.1177/1534735421990080. PMID 33588610
- [Background] Samuels N, Ben-Arye E. Integrative Approaches to Chemotherapy-Induced Peripheral Neuropathy. Curr Oncol Rep. 2020 Feb 11;22(3):23. doi: 10.1007/s11912-020-0891-2. PMID 32048067
- [Background] Ben-Arye E, Dahly H, Keshet Y, Dagash J, Samuels N. Providing integrative care in the pre-chemotherapy setting: a pragmatic controlled patient-centered trial with implications for supportive cancer care. J Cancer Res Clin Oncol. 2018 Sep;144(9):1825-1833. doi: 10.1007/s00432-018-2700-y. Epub 2018 Jul 6. PMID 29980837